CLINICAL TRIAL: NCT06543394
Title: Optimizing Recruitment Methodology for Medication Adherence Interventions: The ENGaging Patients in Adherence Interventions UsinG Behavioral SciencE (ENGAGE) Randomized Factorial Trial
Brief Title: Engaging Patients in Adherence Interventions Using Behavioral Science
Acronym: ENGAGE-HTN
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ian Kronish, Associate Professor of Medicine, Columbia University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: AAAV0521; P30AG064198 (NIH)
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Uncontrolled Hypertension
Keywords: medication adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: PIs and data analysts will be masked to group assignment when analyzing data to determine the effectiveness of the recruitment strategy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Postcard/behavioral letter/4 calls (Active Comparator): Mailed a priming postcard, followed by a prospect theory-informed recruitment letter, followed by up to 4 phone call attempts to schedule patient to attend an adherence counseling session with a clinical pharmacist trained in brief negotiated interviewing
  Interventions: Behavioral: Primer postcard; Behavioral: Behavioral theory-informed recruitment letter; Behavioral: 4 phone calls
- No postcard/behavioral letter/4 calls (Active Comparator): Mailed a prospect-theory informed recruitment letter that is not preceded by a priming postcard, followed by up to 4 phone call attempts to schedule patient to attend an adherence counseling session with a clinical pharmacist trained in brief negotiated interviewing
  Interventions: Behavioral: Behavioral theory-informed recruitment letter; Behavioral: 4 phone calls
- Postcard/control letter/4 calls (Active Comparator): Mailed a priming postcard, followed by a usual care control recruitment letter, followed by up to 4 phone call attempts to schedule patient to attend an adherence counseling session with a clinical pharmacist trained in brief negotiated interviewing
  Interventions: Behavioral: Primer postcard; Behavioral: Control recruitment letter; Behavioral: 4 phone calls
- No postcard/control letter/4 calls (Active Comparator): Mailed a usual care control recruitment letter that is not preceded by a priming postcard, followed by up to 4 phone call attempts to schedule patient to attend an adherence counseling session with a clinical pharmacist trained in brief negotiated interviewing
  Interventions: Behavioral: Control recruitment letter; Behavioral: 4 phone calls
- Postcard/behavioral letter/2 calls (Active Comparator): Mailed a priming postcard, followed by a prospect theory-informed recruitment letter, followed by up to 2 phone call attempts to schedule patient to attend an adherence counseling session with a clinical pharmacist trained in brief negotiated interviewing
  Interventions: Behavioral: Primer postcard; Behavioral: Behavioral theory-informed recruitment letter; Behavioral: 2 phone calls
- No postcard/behavioral letter/2 calls (Active Comparator): Mailed a prospect theory-informed recruitment letter that is not preceded by a priming postcard, followed by up to 2 phone call attempts to schedule patient to attend an adherence counseling session with a clinical pharmacist trained in brief negotiated interviewing
  Interventions: Behavioral: Behavioral theory-informed recruitment letter; Behavioral: 2 phone calls
- Postcard/control letter/2 calls (Active Comparator): Mailed a priming postcard, followed by a usual care control recruitment letter, followed by up to 2 phone call attempts to schedule patient to attend an adherence counseling session with a clinical pharmacist trained in brief negotiated interviewing
  Interventions: Behavioral: Primer postcard; Behavioral: Control recruitment letter; Behavioral: 2 phone calls
- No postcare/control letter/2 calls (Active Comparator): Mailed a usual care control recruitment letter that is not preceded by a priming postcard, followed by up to 2 phone call attempts to schedule patient to attend an adherence counseling session with a clinical pharmacist trained in brief negotiated interviewing
  Interventions: Behavioral: Control recruitment letter; Behavioral: 2 phone calls

INTERVENTIONS:
Behavioral: Primer postcard — Mailed primer postcard
  Arms: Postcard/behavioral letter/2 calls; Postcard/behavioral letter/4 calls; Postcard/control letter/2 calls; Postcard/control letter/4 calls
Behavioral: Control recruitment letter — Mailed recruitment letter with usual care message framing
  Arms: No postcard/control letter/4 calls; No postcare/control letter/2 calls; Postcard/control letter/2 calls; Postcard/control letter/4 calls
Behavioral: Behavioral theory-informed recruitment letter — Mailed recruitment letter with prospect-theory informed message framing
  Arms: No postcard/behavioral letter/2 calls; No postcard/behavioral letter/4 calls; Postcard/behavioral letter/2 calls; Postcard/behavioral letter/4 calls
Behavioral: 2 phone calls — Up to 2 phone call attempts to schedule patient for a clinical pharmacist adherence counseling visit
  Arms: No postcard/behavioral letter/2 calls; No postcare/control letter/2 calls; Postcard/behavioral letter/2 calls; Postcard/control letter/2 calls
Behavioral: 4 phone calls — Up to 4 phone call attempts to schedule patient for a clinical pharmacist adherence counseling visit
  Arms: No postcard/behavioral letter/4 calls; No postcard/control letter/4 calls; Postcard/behavioral letter/4 calls; Postcard/control letter/4 calls

SUMMARY:
The overarching goal of the proposed research is to prepare an evidence-based clinical pharmacist-delivered medication adherence intervention for sustainable implementation and dissemination. Because the effectiveness of the intervention has already been demonstrated in a NIH Stage Model Stage 4 trial called STIC2IT, this study will include an NIH Stage Model Stage 5 Effectiveness-Implementation Type 3 Hybrid design, in which the primary focus is on testing different implementation methods, while secondarily observing clinical effects. The overarching hypothesis is that investigators can identify the most impactful elements of a behavioral theory-informed recruitment approach, which can be replicable across clinical settings.

Accordingly, this study will perform testing of behaviorally-informed recruitment approaches in a primary care setting that serves patients from under-resourced communities. Patients will be English or Spanish speaking adults ≥18 years of age identified through the electronic health record (EHR) as having a primary care clinician at the participating practice as well as uncontrolled hypertension and suboptimal adherence to blood pressure medications based on pharmacy fill data linked to the electronic health record (EHR). The primary care clinicians of eligible patients identified through the EHR will have the opportunity to opt-out any patients they wish not to be included. Patients will then be randomized to each of the following conditions, such that there will be 8 total arms: (1) inclusion of a mailer primer (yes/no), (2) the most successful recruitment letter from a preliminary study using prospect theory (versus the control letter), and (3) intensity of the intervention outreach (up to 4 calls vs. up to 2 calls).

Patients across all arms who agree to be scheduled will receive an appointment with one of the clinical pharmacists trained in the brief negotiated interviewing approach used in the STIC2IT trial. The primary outcome will be completion of a clinical pharmacist appointment within 12 weeks of randomization. Key secondary outcomes will include scheduled visit rates, no-show rates for scheduled appointments, pharmacy fill adherence to statins and blood pressure medications over the 3-month follow-up, and clinical outcomes, including blood pressure as per EHR data in the 3 months after randomization.

DETAILED DESCRIPTION:
Participants will be recruited from Columbia University Irving Medical Center (CUIMC)-affiliated primary care clinics that are part of the New York Presbyterian (NYP) Ambulatory Care Network (ACN). These clinics provide care to patients in the catchment area of CUIMC which is notable for substantial racial, ethnic, and economic diversity. The study team will identify participants with uncontrolled hypertension (last office BP <140/90 mmHg) who also are nonadherent (PDC<80%) to at least one antihypertensive medication class and meet other study eligibility criteria.

Participants will then be randomized using a 2^3 factorial approach to each of the following conditions, such that there will be 8 total arms: (1) inclusion of a mailer primer (yes vs no), (2) a behavioral theory-informed letter script (vs usual scripted letter), and (3) intensity of the recruitment outreach (up to 4 calls vs up to 2 calls). Recruitment outreach will be conducted by members of the study team, who will be trained to deliver different interventions based on a patient's assigned arm. Enrollment will be staggered over an approximately 4-month period so as not to overwhelm the scheduling staff and mimic how quality improvement programs are conducted in typical practice.

Participants who agree to participate in the adherence counseling session after receiving any of the 8 combinations of recruitment strategies will be scheduled to receive a brief evidence-based medication adherence counseling session known as brief negotiated interviewing. Patients who schedule a counseling session with a clinical pharmacist will receive a reminder call before their appointment. This will involve a 30-minute or less telephone or video visit with a nurse or clinical pharmacist who will use a semi-structured guide to confirm the patient's treatment regimen, engage them in sharing potential barriers to adherence or other factors that may be contributing to poor disease control, discuss their readiness to modify behaviors, and work with the patient to develop a shared plan.

The study will concurrently test whether 1) inclusion of a mailed primer is better than no inclusion, 2) whether use of a behavioral theory-informed message-framing strategy in the recruitment letter is better than the usual approach that does not include theory-informed message framing in a recruitment letter, and 3) whether increasing the intensity of recruitment outreach after the letter through up to 4 phone calls is better than up to 2 phone calls. The primary outcome for the study will be whether or not patients completed the adherence counseling session within 12 weeks of randomization. The secondary outcome will be whether patients agreed to have the counseling session scheduled. Exploratory outcomes will include the effects on medication adherence, blood pressure, and LDL cholesterol 3 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Receive care at a Columbia-affiliated primary care clinic in the Ambulatory Care Network
* Diagnosis of hypertension
* Office BP >=140/90 mmHg at most recent office visit
* Prescribed at least one blood pressure medication
* Nonadherent to at least one blood pressure medication as per pharmacy dispense records (proportion of days covered <80% to at least one eligible medication in last 6 months)

Exclusion Criteria:

* Do not speak English or Spanish
* Pregnancy, dementia or terminal conditions as per ICD-10 codes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who completed an adherence counseling session | 12 weeks
  Measures patient attendance at a single adherence counseling session

SECONDARY OUTCOMES:
Number of participants who scheduled an adherence counseling session | 12 weeks
  Patient scheduled an adherence counseling session
Number of days that participants were adherent to blood pressure medication | 12 weeks
  Number of days covered for blood pressure medications >= 80%
Number of days that participants were adherent to statin medication | 12 weeks
  Number of days covered for statin medications >= 80%
Systolic blood pressure | 12 weeks
  Systolic blood pressure at office visit
Diastolic blood pressure | 12 weeks
  Diastolic blood pressure at office visit

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to make available a de-identified database upon request
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Within 1 year of completion of the trial